CLINICAL TRIAL: NCT03199599
Title: Prognostic Positron Emission Tomography/Computed Tomogrpahy Model in Non Small Cell Lung Cancer
Brief Title: Prognostic PET/CT Model in Non Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PRINCE; PRT-K15-119 (Other Grant/Funding Number: INCA)
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: PET/CT; image processing; outcome
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective validation of a prognostic model based on advanced PET/CT image analysis in non small cell lung cancer

DETAILED DESCRIPTION:
Validation on a prospective cohort of patient of a predictive model for survival based on image derived parameters

ELIGIBILITY:
Inclusion Criteria:

* non small cell lung cancer
* initial fluorodeoxygluoces (FDG) PET/CT before treatment

exclusion criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with Non small cell lung cancer undergoing initial staging FDG PET/CT
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
validation of a multiparametric PET/CT prognostic model | 18 months
  overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: MATHIEU HATT, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Chu Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided